CLINICAL TRIAL: NCT02396966
Title: A Prospective, Non-interventional, Observational, Multi-centre Study to Document QoL of Subjects With Acromegaly Under Lanreotide Autogel® Treatment.
Brief Title: Quality of Life (QoL) in Subjects With Acromegaly Under Lanreotide Autogel® Treatment.
Acronym: ACRO QLQ
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-38-52030-306
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the protocol is to evaluate and describe QoL, in the population of Polish acromegalic patients treated with Lanreotide Autogel® 120 mg during the 24 months (long term observation).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with acromegaly treated for at least three months and no longer than three years with Lanreotide Autogel® 120 mg just before inclusion.
* Patients capable of giving their informed consent to participate in the study and who agree to participate by signing the informed consent form.

Exclusion Criteria:

* Active participation in any interventional or any other non-interventional acromegaly clinical study. (Previous participation in any interventional or any observational / post marketing study (PMS) of other somatostatin analogue should not be an exclusion criteria).
* Any medical or psychological condition, according to investigator judgement, that might compromise the ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Specialist care clinic and hospital clinic.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2014-12; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Acromegaly quality of life (AcroQol) questionnaire | Change from baseline (visit 1), visit 3 and 6 (visits occur approximately every 4-5 months, during 2 years of observation)
  The AcroQol questionnaire and total AcroQol score will be analysed descriptively overall and according to hormonal control, presence of prior radiotherapy, presence of prior surgery.

SECONDARY OUTCOMES:
Hormonal control of serum growth hormone (GH) and insulin-like growth factor 1 (IGF-1) concentration | Visit 1 to 6 (visits occur approximately every 4-5 months, during 2 years of observation)
  Descriptive analysis
Clinical symptoms of acromegaly | Visit 1 to 6 (visits occur approximately every 4-5 months, during 2 years of observation)
  Descriptive analysis of the following symptoms - Headache, Sweating, Joint symptoms and Swelling
Patient overall assessment of satisfaction from treatment | Visit 1 to 6 (visits occur approximately every 4-5 months, during 2 years of observation)
  Using a Likert scale (from 1 to 5); completely satisfied, rather satisfied, neither satisfied nor dissatisfied, rather dissatisfied, completely dissatisfied.
Lanreotide injection interval (28, 42 or 56 days) | Visit 1 to 6 (visits occur approximately every 4-5 months, during 2 years of observation)
  Summary of overall and by hormone control status.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (18):
- Poland (18):
  - Bialystok
  - Bydgoszcz
  - Bytom
  - Gdansk
  - Gliwice
  - Katowice
  - Kielce
  - Krakow
  - Lodz
  - Lublin
  - Olsztyn
  - Opole
  - Poznan
  - Rybnik
  - Rzeszów
  - Szczecin
  - Warsaw
  - Wroclaw